CLINICAL TRIAL: NCT01528254
Title: A 5-year Study to Compare the Durability of Glycemic Control of a Combination Regimen With Vildagliptin & Metformin Versus Standard-of-care Monotherapy With Metformin, Initiated in Treatment-naïve Patients With Type 2 Diabetes Mellitus
Brief Title: VERIFY:A Study to Compare Combination Regimen With Vildagliptin & Metformin Versus Metformin in Treatment-naïve Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A23156; 2011-003712-23 (EudraCT Number)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Vildagliptin; Elderly Patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vilda 50mg bid + metformin (Active Comparator): Metformin + vildagliptin
  Interventions: Drug: vildagliptin; Drug: Metformin
- Placebo + metformin (Experimental): Metformin + Placebo of vildagliptin
  Interventions: Drug: Placebo of vildagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Placebo of vildagliptin
  Other Names: Placebo
  Arms: Placebo + metformin
Drug: vildagliptin — One tablet (50 mg oral) of vildagliptin in the morning and one tablet in the evening with or without food.
  Other Names: LAF237
  Arms: Vilda 50mg bid + metformin
Drug: Metformin — Twice daily (bid) regimen during or after meals at the same time as vildagliptin.

SUMMARY:
The purpose of this study was to determine whether the initiation of a vildagliptin plus metformin combination regimen would result in more durable glycemic control than metformin monotherapy in treatment-naïve patients with type-2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This was a multi-center, double-blind, placebo-controlled, 2-arm, parallel group study with a run-in period and up to 5 years treatment period. Following a screening visit (Visit 1) and a screening period of up to 2 weeks, treatment-naïve patients, meeting all eligibility criteria entered the run-in period at Visit 2.

* Run-in period: At Visit 2, in all eligible patients, metformin treatment was initiated and/or up-titrated. At the end of the 3-week run-in period, patients who were able to tolerate a total dose of at least 1000 mg and up to 2000 mg daily proceeded to randomization and started in Period 1.
* Period 1 (vildagliptin/metformin combination versus metformin): At Visit 3, patients were randomized 1:1 to one of the following study regimens:

  * Metformin up to 1000 mg bid plus vildagliptin 50mg bid or
  * Metformin up to 1000 mg bid plus matching placebo bid

The duration of Period 1 could differ between patients depending on the time when the second of two HbA1c measurements taken at two consecutive visits after randomisation confirmed HbA1c ≥ 7.0%.

• Period 2 (vildagliptin/metformin combination versus vildagliptin add-on to metformin): In the case of two consecutive HbA1c measurements ≥7.0% from two consecutive study visits during Period 1, patients who were randomised to the placebo arm in Period 1 received vildagliptin 50 mg bid. Patients who were randomised to the active vildagliptin 50 mg bid arm in Period 1 continued to receive vildagliptin 50 mg bid. All patients continued to take their metformin dose unchanged. Period 2 remained masked to the patient and both patients and investigators remained masked to the treatment allocation in Period 1.

If, during Period 2, therapy intensification was required in accordance with the local guidelines, the patient entered Period 3. The duration of Period 2 could differ between patients. End of Period 2 was considered when insulin treatment was initiated, or alternatively when the patient was discontinued because insulin treatment was not initiated in Period 3.

• Period 3 (insulin initiation): In Period 3, patients were to be initiated on open-label insulin. The study drug regimen continued unchanged and remained masked to the patient in Period 3 and both patients and investigators remained masked to the treatment allocation in Period 1.

ELIGIBILITY:
Key Inclusion Criteria:

* Type 2 Diabetes Mellitus (T2DM) diagnosed ≤ 24 months ago
* glycosylated hemoglobin (HbA1c) ≥6.5% and ≤7.5% at Visit 1
* Treatment-naïve.
* Body mass index (BMI) ≥22 and ≤40 kg/m2 at Visit 1

Key Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Fasting plasma glucose (FPG) ≥ 270 mg/dL (≥ 15.0 mmol/L)
* Previous or current participation in any vildagliptin clinical study.
* History of hypersensitivity to dipeptidyl peptidase-4 (DPP-4) inhibitors.
* Concurrent medical condition that may interfere with the interpretation of efficacy and safety data during the study.
* Donation of blood or significant blood loss equaling to at least one unit of blood within the past 2 weeks of start of study or a blood transfusion within the past 12 weeks or planned regular transfusions during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2012-03-30 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (188):
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
- Australia (3):
  - Novartis Investigative Site, Brookvale, New South Wales
  - Novartis Investigative Site, Woy Woy, New South Wales
  - Novartis Investigative Site, Morayfield, Queensland
- Novartis Investigative Site, Vienna, Austria
- Brazil (8):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Mogi das Cruzes, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (7):
  - Novartis Investigative Site, Smolyan, Bulgaria
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Kazanlak
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Razgrad
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
- Colombia (4):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Baranquilla
  - Novartis Investigative Site, Bogotá
- Czechia (4):
  - Novartis Investigative Site, Písek, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brandýs nad Labem
  - Novartis Investigative Site, Prague
- Dominican Republic (2):
  - Novartis Investigative Site, Santo Domingo, Republica Dominicana
  - Novartis Investigative Site, Santo Domingo
- Estonia (2):
  - Novartis Investigative Site, Saku
  - Novartis Investigative Site, Tallinn
- Finland (4):
  - Novartis Investigative Site, Lahti, Suomi
  - Novartis Investigative Site, Kerava
  - Novartis Investigative Site, Kouvola
  - Novartis Investigative Site, Tampere
- Germany (14):
  - Novartis Investigative Site, Hainstadt, Hainburg
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Kamp-Lintfort
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Saint Ingbert - Oberwuerzbach
  - Novartis Investigative Site, Wangen
- Guatemala (2):
  - Novartis Investigative Site, Clinica, Departamento de Guatemala
  - Novartis Investigative Site, Guatemala City
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (7):
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Csongrád
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Kalocsa
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
- India (8):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Indore, Madhya Pradesh
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Chandigarh
- Israel (7):
  - Novartis Investigative Site, Haifa, Israel
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Sefad
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Giborim, Holon
- Italy (6):
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Campobasso, CB
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Roma, RM
- Latvia (7):
  - Novartis Investigative Site, Jelgava, LV
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Ogre, LV
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Talsi, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lithuania (5):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Jonava
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Vilnius
- Malaysia (2):
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (7):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Cuautla, Morelos
  - Novartis Investigative Site, Cuernavaca, Morelos
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Distrito Federal
  - Novartis Investigative Site, Durango
  - Novartis Investigative Site, Querétaro
- Norway (5):
  - Novartis Investigative Site, Enebakk
  - Novartis Investigative Site, Fetsund
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Spikkestad
- Novartis Investigative Site, Panama City, Panama
- Peru (7):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, Chorrillos, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Magdalena, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Arequipa
- Philippines (6):
  - Novartis Investigative Site, Marikina City, National Capital Region
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Pasay, Philippines
  - Novartis Investigative Site, Marikina City
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, San Juan City
- Poland (3):
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Romania (5):
  - Novartis Investigative Site, Oradea, Bihor County
  - Novartis Investigative Site, Oradea, Jud. Bihor
  - Novartis Investigative Site, Ploieşti, Jud. Prahova
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Timișoara
- Russia (8):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
- Slovakia (17):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Lučenec, Slovak Republic
  - Novartis Investigative Site, Námestovo, Slovak Republic
  - Novartis Investigative Site, Rožňava, Slovak Republic
  - Novartis Investigative Site, Šaľa, Slovak Republic
  - Novartis Investigative Site, Trebišov, Slovak Republic
  - Novartis Investigative Site, Žilina, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Sabinov
  - Novartis Investigative Site, Sereď
  - Novartis Investigative Site, Štúrovo
  - Novartis Investigative Site, Žilina
- South Africa (6):
  - Novartis Investigative Site, Alberton
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, Gauteng
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Pretoria
- South Korea (8):
  - Novartis Investigative Site, Incheon, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Daejeon
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Sant Adria Del Besos, Barcelona
  - Novartis Investigative Site, Santa Coloma de Gramanet, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
- Taiwan (4):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Xindian District
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Diskapi / Ankara, Turkey
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Denizli
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tsotra F, Kappel M, Peristeris P, Bader G, Levi E, Lister N, Malhotra A, Ostwald DA. The societal impact of early intensified treatment in patients with type 2 diabetes mellitus. J Comp Eff Res. 2022 Nov;11(16):1185-1199. doi: 10.2217/cer-2022-0110. Epub 2022 Sep 28. PMID 36170017
- [Derived] Vencio S, Manosalva JP, Mathieu C, Proot P, Lozno HY, Paldanius PM. Exploring early combination strategy in Latin American patients with newly diagnosed type 2 diabetes: a sub-analysis of the VERIFY study. Diabetol Metab Syndr. 2021 Jun 15;13(1):68. doi: 10.1186/s13098-021-00686-9. PMID 34130731
- [Derived] Matthews D, Del Prato S, Mohan V, Mathieu C, Vencio S, Chan JCN, Stumvoll M, Paldanius PM. Insights from VERIFY: Early Combination Therapy Provides Better Glycaemic Durability Than a Stepwise Approach in Newly Diagnosed Type 2 Diabetes. Diabetes Ther. 2020 Nov;11(11):2465-2476. doi: 10.1007/s13300-020-00926-7. Epub 2020 Sep 25. PMID 32975711
- [Derived] Matthews DR, Paldanius PM, Proot P, Chiang Y, Stumvoll M, Del Prato S; VERIFY study group. Glycaemic durability of an early combination therapy with vildagliptin and metformin versus sequential metformin monotherapy in newly diagnosed type 2 diabetes (VERIFY): a 5-year, multicentre, randomised, double-blind trial. Lancet. 2019 Oct 26;394(10208):1519-1529. doi: 10.1016/S0140-6736(19)32131-2. Epub 2019 Sep 18. PMID 31542292
- [Derived] Matthews DR, Paldanius PM, Proot P, Foley JE, Stumvoll M, Del Prato S. Baseline characteristics in the VERIFY study: a randomized trial assessing the durability of glycaemic control with early vildagliptin-metformin combination in newly diagnosed Type 2 diabetes. Diabet Med. 2019 Apr;36(4):505-513. doi: 10.1111/dme.13886. Epub 2019 Feb 12. PMID 30576013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to screen approximately 4000 patients in order to randomize 2000 patients. Actually, 2001 patients were randomized, 998 patients into the Vilda 50mg bid + metformin group and 1003 into the placebo + metformin group.
Groups:
- Vilda 50mg Bid + Metformin: vildagliptin (Vilda 50mg bid) + Metformin
- Placebo + Metformin: Placebo of vildagliptin (Vilda 50mg bid) + Metformin
Period: Overall Study
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Started (All randomized patients (RAN)) | 998 | 1003
Safety Set (At least one dose of study medication) | 998 | 1001
Full Analysis Set (FAS) (At least one randomized study medication and a post-randomization efficacy parameter assessment.) | 983 | 989
Completed Treatment Period 1 | 458 | 273
Completed Treatment Period 2 | 244 | 399
Completed Treatment Period 3 | 109 | 115
Completed | 811 | 787
Not Completed | 187 | 216
Not completed — Administrative problems | 96 | 94
Not completed — Adverse Event | 28 | 44
Not completed — Lost to Follow-up | 17 | 24
Not completed — Death | 13 | 9
Not completed — Protocol deviation | 9 | 19
Not completed — New therapy for study indication | 8 | 6
Not completed — Unsatisfactory therapeutic effect | 6 | 8
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Abnormal laboratory value(s) | 3 | 7
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — No longer requires study drug | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin | Total
Number analyzed (Participants) | 998 | 1003 | 2001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (9.54) | 54.6 (9.24) | 54.3 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 545 | 515 | 1060
  Male | 453 | 488 | 941
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 605 | 612 | 1217
  Black | 26 | 23 | 49
  Asian | 186 | 187 | 373
  Native American | 103 | 107 | 210
  Other | 78 | 74 | 152
glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent] — Baseline HbA1c is the sample obtained on day 1, or the sample obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurement is missing. Population: Only patients with at least one measurement on or prior to Day 1 are included.
  Percent
    number analyzed (Participants) | 996 | 1003 | 1999
    (all) | 6.7 (0.45) | 6.7 (0.47) | 6.7 (0.46)
fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/l] — Baseline FPG is the sample obtained on day 1, or the sample obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurement is missing. Population: Only patients with at least one measurement on or prior to Day 1 are included.
  mmol/l
    number analyzed (Participants) | 996 | 1003 | 1999
    (all) | 7.1 (1.40) | 7.2 (1.47) | 7.1 (1.44)
Duration of type 2 diabetes [Mean (Standard Deviation); unit: months] — Duration of type 2 diabetes is collected on the day of the screening measurement (Week -5, Visit 1)
  months | 6.2 (7.00) | 6.6 (8.05) | 6.4 (7.55)
Glomerular Filtration Rate (Modification of Diet in Renal Disease) [Count of Participants; unit: Participants] — GFR (MDRD) = GFR estimated using the MDRD formula. Baseline GFR is calculated using the serum creatinine and body weight value at the Day 1 measurement, or the value obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurement is missing. Age is the value at screening.
  Participants
    Normal (>80) | 660 | 661 | 1321
    Mild (>=50 - <=80) | 333 | 337 | 670
    Moderate (>=30 - <50) | 3 | 4 | 7
    Severe (<30) | 0 | 1 | 1
    Missing | 2 | 0 | 2
Is subject a current smoker? [Count of Participants; unit: Participants] — Smoking status is collected on the day of the screening measurement (Week -5, Visit 1)
  Participants
    Is subject a current smoker?=Yes | 154 | 136 | 290
    Is subject a current smoker?=No | 844 | 867 | 1711

OUTCOME MEASURES:

1. Primary Outcome: Time to Initial Treatment Failure
Description: Treatment failure was defined as two consecutive scheduled visits with HbA1c >= 7.0% (starting from 13 weeks after randomization) and the time to treatment failure was the number of days from randomization to the second of the consecutive scheduled visits.
  Participants who discontinued the study for any reason during Period 1 were censored at the date of discontinuation. Participants who remained under the threshold (or whose measurement above the threshold was not confirmed at next scheduled visit) were censored at the date of last study visit.
Time Frame: Visit 4 (Week 13) up to End of Study (Study Drug Discontinuation or Premature Subject Discontinuation)
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 983 | 989
Rate (%)
  Weeks 13-52: number analyzed (Participants) | 75 | 192
  Weeks 13-52 | 7.81 [6.28 to 9.70] | 19.97 [17.58 to 22.65]
  Year 2: number analyzed (Participants) | 168 | 326
  Year 2 | 17.79 [15.49 to 20.38] | 34.67 [31.72 to 37.82]
  Year 3: number analyzed (Participants) | 290 | 446
  Year 3 | 31.24 [28.35 to 34.33] | 48.31 [45.12 to 51.61]
  Year 4: number analyzed (Participants) | 365 | 540
  Year 4 | 39.84 [36.74 to 43.11] | 59.29 [56.08 to 62.53]
  Year 5: number analyzed (Participants) | 421 | 600
  Year 5 | 46.41 [43.20 to 49.74] | 66.57 [63.43 to 69.69]
  > Year 5: number analyzed (Participants) | 429 | 614
  > Year 5 | 52.67 [44.29 to 61.58] | 74.39 [68.39 to 80.04]
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.45 to 0.58]

2. Secondary Outcome: Rate of Loss in Glycemic Control During Period 1
Description: The rate of loss in glycemic control was estimated using the slope of HbA1c over time (years).
  HbA1c data collected from Week 26 up to and including the end of Period 1 visit was included in the analysis. Baseline HbA1c was the sample obtained on day 1, or the sample obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurement was missing. End of Period 1 was defined as the final post-baseline assessment obtained at any visit within Period 1 (scheduled or unscheduled), up to the last scheduled visit.
Time Frame: Visit 5 (Week 26) to End of Period 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 983 | 989
Rate (%) | 0.24 (0.01) | 0.27 (0.01)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; Test type: Other; p = 0.042, Mixed Models Analysis; Slope = -0.02, 95% CI 2-sided [-0.05 to 0.00], Standard Error of Mean 0.01

3. Secondary Outcome: Rate of Loss in Glycemic Control in HbA1c Over Time During Period 2
Description: The rate of loss in glycemic control was estimated using the slope of HbA1c over time (years).
  HbA1c data collected from 26 weeks after the start of Period 2 to the end of Period 2 were included in the analysis, for participants who started insulin therapy in Period 3 or discontinued during Period 2 due to being unable or unwilling to initiate insulin therapy in period 3. Participants who completed the study in Period 1 or Period 2 were not be included in the analysis.
Time Frame: From 26 weeks after start of Period 2 to end of Period 2
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 410 | 588
Rate (%) | 1.11 (0.15) | 1.02 (0.12)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; Test type: Other; p = 0.635, Mixed Models Analysis; Slope = 0.09, 95% CI 2-sided [-0.29 to 0.47], Standard Error of Mean 0.19

4. Secondary Outcome: Rate of Loss in Glycemic Control in Fasting Plasma Glucose (FPG) During Period 1
Description: Rate of loss in glycemic control was estimated using the slope of FPG over time (years).
  FPG (fasting plasma glucose) data from Week 26 to the end of Period 1 was included in the analysis. Baseline FPG was the sample obtained on day 1, or the sample obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurement is missing. Participants who completed the study in Period 1 or Period 2 were not be included in the analysis.
Time Frame: Visit 5 (Week 26) to End of Period 1
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 983 | 989
Rate (%) | 0.25 (0.01) | 0.26 (0.01)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; Test type: Other; p = 0.530, Mixed Models Analysis; Slope = -0.01, 95% CI 2-sided [-0.05 to 0.02], Standard Error of Mean 0.02

5. Secondary Outcome: Rate of Loss in Glycemic Control in Fasting Plasma Glucose (FPG) Over Time During Period 2
Description: Rate of loss in glycemic control was estimated using the slope of FPG over time (years).
  FPG (fasting plasma glucose) data from 26 weeks after the start of Period 2 to then end of Period 2 was included in the analysis. Only participants who started insulin therapy in Period 3 or discontinued during Period 2 due to being unable or unwilling to initiate insulin therapy in period 3 were included. Participants who completed the study in Period 1 or Period 2 were not be included in the analysis.
Time Frame: From 26 weeks after start of Period 2 to end of Period 2
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 410 | 588
Rate (%) | 1.27 (0.25) | 0.99 (0.19)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; Test type: Other; p = 0.381, Mixed Models Analysis; Slope = 0.28, 95% CI 2-sided [-0.35 to 0.90], Standard Error of Mean 0.32

6. Secondary Outcome: Rate of Loss of Beta Cell Function From Baseline to End of Study
Description: The rate of change of beta cell function was assessed using the slope of AUC of ISR/G over time (years) where AUC of ISR/G is defined as (Area under curve of Insulin secretion rate (derived using c-peptide))/(Area under curve of Glucose), using meal-test data from 0 to 120 minutes. Baseline AUC of ISR/G was derived based on samples obtained on day 1, or samples obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurements were missing. Three analyses were included, using data from Week 13 to the end of Period 1, end of Period 2 and end of study, respectively.
Time Frame: Visit 4 (Week 13), End of Period 1, End of Period 2, End of Study (Study Drug Discontinuation or Premature Subject Discontinuation)
Population: Full Analysis Set (FAS) meal-test subset
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 228 | 227
Rate (%)
  From Week 13 to end of Period 1: number analyzed (Participants) | 201 | 202
  From Week 13 to end of Period 1 | -0.60 (0.15) | -0.53 (0.18)
  From Week 13 to end of Period 2: number analyzed (Participants) | 202 | 204
  From Week 13 to end of Period 2 | -0.93 (0.14) | -0.43 (0.15)
  From Week 13 to end of study: number analyzed (Participants) | 202 | 204
  From Week 13 to end of study | -1.04 (0.15) | -0.46 (0.15)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of Period 1; Test type: Other; p = 0.744, Mixed Models Analysis; Slope = -0.08, 95% CI 2-sided [-0.53 to 0.38], Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of Period 2; Test type: Other; p = 0.017, Mixed Models Analysis; Slope = -0.50, 95% CI 2-sided [-0.91 to -0.09], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of study; Test type: Other; p = 0.006, Mixed Models Analysis; Slope = -0.58, 95% CI 2-sided [-0.99 to -0.17], Standard Error of Mean 0.21

7. Secondary Outcome: Rate of Change in Insulin Sensitivity From Baseline to End of Study
Description: The rate of change of insulin sensitivity is assessed using the slope of OGIS over time (years) where Oral glucose insulin sensitivity (OGIS) was calculated as a function of glucose and insulin, using meal-test data from 0 to 120 minutes. Baseline OGIS is derived based on samples obtained on day 1, or samples obtained at an earlier visit (scheduled or unscheduled) which was closest to Day 1, if the Day 1 measurements are missing. Three analyses were included, using data from Week 13 to the end of Period 1, end of Period 2 and end of study, respectively.
Time Frame: as for outcome 6
Population: Full Analysis Set (FAS) meal-test subset
Measure: Mean (Standard Error); unit: Rate (%)
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 228 | 227
Rate (%)
  From Week 13 to end of Period 1: number analyzed (Participants) | 189 | 193
  From Week 13 to end of Period 1 | -4.61 (1.38) | 0.41 (1.66)
  From Week 13 to end of Period 2: number analyzed (Participants) | 190 | 194
  From Week 13 to end of Period 2 | -6.07 (1.20) | -0.99 (1.24)
  From Week 13 to end of study: number analyzed (Participants) | 190 | 194
  From Week 13 to end of study | -6.39 (1.15) | -1.01 (1.17)
Statistical Analysis 1: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of Period 1; Test type: Other; p = 0.020, Mixed Models Analysis; Slope = -5.03, 95% CI 2-sided [-9.26 to -0.79], Standard Error of Mean 2.16
Statistical Analysis 2: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of Period 2; Test type: Other; p = 0.003, Mixed Models Analysis; Slope = -5.08, 95% CI 2-sided [-8.46 to -1.69], Standard Error of Mean 1.73
Statistical Analysis 3: Comparison: Vilda 50mg Bid + Metformin vs Placebo + Metformin; From Week 13 to end of study; Test type: Other; p = 0.001, Mixed Models Analysis; Slope = -5.38, 95% CI 2-sided [-8.61 to -2.16], Standard Error of Mean 1.64

8. Secondary Outcome: Percentage of Participants With Adverse Events, Serious Adverse Events and Death
Description: Analysis of absolute and relative frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC) in each treatment arm to demonstrate that LAF237 is safe for the treatment of naïve patients with type 2 diabetes mellitus through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: From first dose of study treatment until End of Study (Study Drug Discontinuation or Premature Subject Discontinuation)
Population: Safety Set (SAF). Percentages are based on the number of patients starting each period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin
Number analyzed (Participants) | 998 | 1001
Percentage of Participants
  On-treatment Adverse Event (AEs): number analyzed (Participants) | 833 | 833
  On-treatment Adverse Event (AEs) | 83.5 | 83.2
  On-treatment Serious Adverse Event (SAEs): number analyzed (Participants) | 166 | 183
  On-treatment Serious Adverse Event (SAEs) | 16.6 | 18.3
  On-treatment Deaths: number analyzed (Participants) | 13 | 9
  On-treatment Deaths | 1.3 | 0.9

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 75.6 months.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. Maximum exposure to study treatments = 75.6 months (Vilda 50mg bid + metformin arm) and 66.2 months (Placebo + metformin arm).
Groups:
- Total: Total
Arm/Group | Vilda 50mg Bid + Metformin | Placebo + Metformin | Total
All-Cause Mortality (participants affected / at risk) | 13/998 | 9/1001 | 22/1999
Serious Adverse Events (participants affected / at risk) | 166/998 | 183/1001 | 349/1999
Other Adverse Events (participants affected / at risk) | 582/998 | 566/1001 | 1148/1999
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vilda 50mg Bid + Metformin (N=998) | Placebo + Metformin (N=1001) | Total (N=1999)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 3 | 3
Acute myocardial infarction (Cardiac disorders) | 3 | 4 | 7
Angina pectoris (Cardiac disorders) | 2 | 4 | 6
Angina unstable (Cardiac disorders) | 2 | 1 | 3
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 5 | 11
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 3 | 4 | 7
Cardiac failure acute (Cardiac disorders) | 2 | 1 | 3
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 1
Conduction disorder (Cardiac disorders) | 0 | 2 | 2
Coronary artery disease (Cardiac disorders) | 1 | 3 | 4
Coronary artery insufficiency (Cardiac disorders) | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 3 | 4
Mitral valve disease (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 7 | 10
Myocardial ischaemia (Cardiac disorders) | 2 | 3 | 5
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 2 | 2
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 1
Congenital intestinal malformation (Congenital, familial and genetic disorders) | 0 | 1 | 1
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 1 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Goitre (Endocrine disorders) | 1 | 1 | 2
Hypoparathyroidism (Endocrine disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 2
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 7 | 7
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2 | 2
Rectal prolapse (Gastrointestinal disorders) | 1 | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 4 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 3
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1
Death (General disorders) | 2 | 0 | 2
Granuloma (General disorders) | 0 | 1 | 1
Inflammation (General disorders) | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 1
Peripheral swelling (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 2 | 0 | 2
Stent-graft endoleak (General disorders) | 1 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 2 | 6
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 2 | 5 | 7
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 1
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 2
Appendicitis (Infections and infestations) | 2 | 2 | 4
Bartholin's abscess (Infections and infestations) | 1 | 0 | 1
Bone tuberculosis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Cervicitis (Infections and infestations) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 2 | 1 | 3
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 2
Epididymitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Hepatic echinococciasis (Infections and infestations) | 0 | 1 | 1
Hepatitis viral (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 2
Infection (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 1 | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1 | 1
Pancreas infection (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 14 | 5 | 19
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 1 | 2
Sepsis (Infections and infestations) | 1 | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 3 | 5
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Viral myelitis (Infections and infestations) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 1 | 2
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 1 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 4 | 5
Multiple injuries (Injury, poisoning and procedural complications) | 3 | 0 | 3
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
HIV test positive (Investigations) | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 5 | 7
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 4
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Malignant splenic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oligoastrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 5
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 6
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Refractory cytopenia with multilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3
Brain oedema (Nervous system disorders) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 1 | 3
Cerebral infarction (Nervous system disorders) | 1 | 2 | 3
Cerebral ischaemia (Nervous system disorders) | 0 | 4 | 4
Cerebrovascular accident (Nervous system disorders) | 2 | 2 | 4
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 1
Demyelination (Nervous system disorders) | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 5 | 7
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 2
Radiculopathy (Nervous system disorders) | 2 | 0 | 2
Sciatica (Nervous system disorders) | 3 | 1 | 4
Seizure (Nervous system disorders) | 1 | 1 | 2
Syncope (Nervous system disorders) | 0 | 2 | 2
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Pregnancy with contraceptive device (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Eating disorder (Psychiatric disorders) | 0 | 1 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 2
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 3 | 2 | 5
Renal colic (Renal and urinary disorders) | 1 | 2 | 3
Renal failure (Renal and urinary disorders) | 0 | 3 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Stag horn calculus (Renal and urinary disorders) | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 2
Cervical cyst (Reproductive system and breast disorders) | 0 | 1 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 1
Genital ulceration (Reproductive system and breast disorders) | 0 | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 4 | 5
Ovarian fibrosis (Reproductive system and breast disorders) | 0 | 1 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 2
Haematoma (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 4 | 6
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 1
Peripheral venous disease (Vascular disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 2 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vilda 50mg Bid + Metformin (N=998) | Placebo + Metformin (N=1001) | Total (N=1999)
Diarrhoea (Gastrointestinal disorders) | 104 | 104 | 208
Bronchitis (Infections and infestations) | 58 | 59 | 117
Influenza (Infections and infestations) | 93 | 64 | 157
Nasopharyngitis (Infections and infestations) | 104 | 108 | 212
Upper respiratory tract infection (Infections and infestations) | 83 | 69 | 152
Urinary tract infection (Infections and infestations) | 72 | 69 | 141
Dyslipidaemia (Metabolism and nutrition disorders) | 58 | 71 | 129
Arthralgia (Musculoskeletal and connective tissue disorders) | 100 | 94 | 194
Back pain (Musculoskeletal and connective tissue disorders) | 105 | 86 | 191
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 54 | 40 | 94
Pain in extremity (Musculoskeletal and connective tissue disorders) | 67 | 74 | 141
Dizziness (Nervous system disorders) | 67 | 41 | 108
Headache (Nervous system disorders) | 82 | 72 | 154
Hypertension (Vascular disorders) | 103 | 124 | 227

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01528254/SAP_000.pdf
  • Study Protocol (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT01528254/Prot_001.pdf